CLINICAL TRIAL: NCT06475781
Title: A Multinational Phase 2, Randomized, Double-Blinded, Placebo-Controlled, Multiple-Dose Study to Evaluate the Safety and Efficacy of Mirivadelgat, an Aldehyde Dehydrogenase 2 Activator, in Patients With Pulmonary Hypertension Associated With Interstitial Lung Disease (PH-ILD)
Brief Title: Study to Evaluate Safety and Efficacy of Mirivadelgat in PH-ILD
Acronym: WINDWARD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Collaborators: QPS-Qualitix Clinical Research Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FP-045C-23-001
Record Dates: First submitted 2024-06-12; First posted 2024-06-26 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Group 3 Pulmonary Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blinded, Placebo-Controlled, Multiple-Dose Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug will be provided in wallet cards. The wallet cards will have unique numbering and will be assigned by an interactive web response system (IWRS). The capsules containing active drug and the placebo capsules will have the same appearance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 150 mg mirivadelgat (Experimental): 150 mg mirivadelgat once daily
  Interventions: Drug: Mirivadelgat
- 300 mg mirivadelgat (Experimental): 300 mg mirivadelgat once daily
  Interventions: Drug: Mirivadelgat
- placebo (Placebo Comparator): placebo once daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mirivadelgat — Selective aldehyde dehydrogenase 2 (ALDH2) activator
  Other Names: FP-045
  Arms: 150 mg mirivadelgat; 300 mg mirivadelgat
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to see if mirivadelgat will work in patients with Pulmonary Hypertension Associated with Interstitial Lung Disease (PH-ILD). It will also learn about the safety of mirivadelgat. The main question it aims to answer is if mirivadelgat will improve pulmonary vascular resistance (PVR). Pulmonary vascular resistance is a way to measure blood flow in the lungs.

Researchers will compare mirivadelgat to a placebo (a look-alike capsule that contains no drug) to see if mirivadelgat works to improve the symptoms of PH-ILD. The symptoms of PH-ILD that are being looked at are exercise tolerance, heart function, and general well-being.

Participants will:

Take mirivadelgat or a placebo once a day for 12 weeks

Visit the clinic once every 4 weeks for checkups and tests

Receive phone calls every one or two weeks to check on how things are going

DETAILED DESCRIPTION:
The study is a phase 2, multinational, double-blind, 3-arm study to evaluate the safety and efficacy of mirivadelgat, an aldehyde dehydrogenase 2 activator, in adult subjects (aged 18 to 85 years) with PH-ILD. Subjects must have a confirmed diagnosis of ILD as defined by the American Thoracic Society (ATS), European Respiratory Society (ERS), Japanese Respiratory Society (JRS), and/or Latin American Thoracic Society (ALAT) guidelines (Raghu, 2018). The diagnosis is based on a HRCT either performed at screening or within 180 days prior to screening or a historical surgical biopsy (or other appropriate tissue sampling (e.g., cryobiopsy)) and an RHC performed at screening. Subjects who also have connective tissue disorders can comprise up to 20% of the study population.

To be eligible for the study, a subject must be willing to undergo a Right Heart Catheterization (RHC) during screening and at the Week 12 Visit (at the end of study treatment). Subjects on chronic treatment for underlying pulmonary diseases must be on a stable/optimized dose for ≥30 days prior to screening and have been receiving treatment for ≥90 days prior to screening.

The study will enroll approximately 126 subjects, assuming a drop-out rate of 20%, to obtain 99 evaluable subjects (33 evaluable subjects in each cohort).

Study visits will include a Screening Visit; Visit 2 (Study Day 1); Weeks 2, 3, 4, 6, 8,10, and 12 Visits (+/ 3 days); and a safety Follow-up Visit (+/ 3 days) after the Week 12 Visit. Visits on Weeks 2, 3, 6, and 10 will be conducted by phone calls.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of PH-ILD.
2. Subject voluntarily gives informed consent.
3. Subjects aged between 18 and 85 years at the time of signing informed consent.
4. Subjects must agree to practice protocol-defined birth control during the study period.

   * Males with a partner of childbearing potential must practice protocol-defined birth control for the duration of treatment and at least 96 hours after discontinuing the IP.
   * Female subjects of childbearing of potential (including those <1-year post menopausal) must practice protocol-defined birth control during the conduct of the study and for 30 days after the last dose of IP (males only during exposure to IP).
   * Women not of childbearing potential are defined as:

     1. Post-menopausal women (at least 12 months with no menses without an alternative medical cause); in women <45 years of age, a high follicle-stimulating hormone (FSH) level in the post-menopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy; OR
     2. Have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion, at least 6 weeks prior to screening; OR
     3. Have a congenital or acquired condition that prevents childbearing.
5. The subject has a confirmed diagnosis of any form of interstitial lung disease based on high resolution computed tomography (HRCT) of the chest within 180 days prior to screening or at screening or a historical surgical biopsy (or other appropriate tissue sampling (e.g., cryobiopsy). The subject can have other findings (e.g., emphysema) if this is not the predominant feature on the scan.
6. Subjects have undergone RHC during the screening period with the following documented parameters:

   * Pulmonary vascular resistance (PVR) ≥4 Wood units and
   * Pulmonary capillary wedge pressure (PCWP) of ≤12 mmHg [if PVR ≥4 Wood units to <6.25 Wood units] or PCWP ≤15 mmHg [if PVR ≥6.25 Wood units] (a left ventricular end diastolic pressure [LVEDP] will be acceptable if a reliable PCWP cannot be obtained) and
   * A mean pulmonary arterial pressure (PAP) of >20 mmHg.
7. Subjects must have a baseline 6-minute walk distance ≥100 meters and ≤500 meters.
8. Subjects agree to a repeat RHC, Chest CT, and MRI prior to study completion.
9. Subjects on chronic treatment for underlying lung disease (i.e., nintedanib or pirfenidone or immunosuppressive agents etc.) must be on a stable/optimized dose for ≥30 days prior to screening and have been receiving treatment for ≥90 days.
10. Subjects on supportive medications (e.g., inhalers for asthma) must be on stable doses for ≥30 days prior to screening.
11. In the Investigator's opinion, the subject must be able to consent for themselves and communicate with local staff using interpreters if necessary. Subjects must agree to attend all study visits and be contactable through a cellular device or landline.
12. Subjects must have clinical laboratory values within normal ranges or <1.5 times the upper limit of normal (ULN) as specified by the testing laboratory.
13. Pulmonary function test (PFT) showing a percent predicted forced vital capacity (FVC) <70% of predicted and diffusion capacity of carbon monoxide (DLCO) <70% corrected for hemoglobin (Hb) value ≥25% and ≤90% at screening (DLCO determined locally must be <70%) using the American Thoracic Society (ATS) standards.
14. Subjects with a prior diagnosis of connective tissue diseases, specifically systemic sclerosis (scleroderma), systemic lupus erythematosus, Sjogren's disease, polymyositis/dermatomyositis/antisynthetase syndrome, rheumatoid arthritis can be included in the study, but no more than 20% of total subjects.
15. Negative serology test for hepatitis B surface antigen and hepatitis C antibody at Screening Visit.

Exclusion Criteria:

Medical Conditions

1. Subject has another concomitant diagnosis of pulmonary hypertension not otherwise considered to be PH-ILD. This would include and is not limited to the concomitant presence of thromboembolic disease, untreated/inadequately treated obstructive sleep apnea, human immunodeficiency virus (HIV), methamphetamine or anorexigenic drug use, and other conditions of the WHO Group 1, 2, 4, and 5 classifications.
2. Subject has evidence of clinically significant left-sided heart disease within 6 months as defined by:

   * Left ventricular ejection fraction <40% as assessed by echocardiography.
   * More than mild left-sided valvulopathy (e.g., worse than mild mitral stenosis or regurgitation and worse than mild aortic stenosis or regurgitation).
   * LVEDP or PCWP >15 mmHg (or >12 mmHg if PVR ≥4 to 6.25 Wood units).
3. Subjects must NOT have 3 or more of the following left ventricular disease/dysfunction risk factors at screening:

   * Body mass index (BMI) ≥30 kg/m2.
   * Uncontrolled diabetes, HbA1C >9.5%, urine glycosuria >1.0 g/dl, or presence of diabetic ketoacidosis
   * History of significant coronary disease within 6 months of screening as demonstrated by any of the following:

     1. History of myocardial infarction or acute coronary syndrome (unstable angina), or
     2. Percutaneous coronary intervention or percutaneous transluminal angioplasty, or previous coronary artery bypass graft, or
     3. Evidence of coronary artery disease (>50% stenosis in at least one major coronary artery) or abnormal nuclear stress test.
4. The subject is receiving >10 L/min of oxygen supplementation by any mode of delivery at rest.
5. The subject has received any PH-approved therapy, including phosphodiesterase type 5 inhibitor, soluble guanylate cyclase inhibitor, endothelin receptor antagonist, or parenteral or oral prostacyclin therapy (excluding vasoreactivity testing) within 60 days of randomization or 5 half-lives. Inhaled prostacyclin (e.g., inhaled treprostinil) on stable doses for ≥30 days prior to screening will be allowed irrespective of local approval (as per ESC/ERS 2022).
6. Use of any potent inhibitors and potent inducers of cytochrome P450 3A4 (CYP3A4) (e.g., boceprevir, cobicistat, danoprevir and ritonavir, elvitegravir and ritonavir, grapefruit juice, indinavir and ritonavir, itraconazole, ketoconazole, lopinavir and ritonavir, paritaprevir and ritonavir and (ombitasvir and/or dasabuvir), posaconazole, ritonavir, saquinavir and ritonavir, telaprevir, tipranavir and ritonavir, telithromycin, troleandomycin, voriconazole, clarithromycin, idelalisib, nefazodone, nelfinavir, carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, St. John's wort).
7. Recent exacerbation of underlying lung disease or active pulmonary/upper respiratory tract infection within 4 weeks of randomization.
8. Any current active malignancy (this does not include localized cancers such as basal or squamous cell carcinoma of the skin). Any history of malignancy that is likely to result in mortality or require significant medical or surgical intervention within the following year.
9. Chronic kidney disease Stage IV or greater (i.e., eGFR ˂30 mL/min/1.73m2) or evidence of acute kidney injury.
10. The subject has a history of congenital heart disease irrespective of any prior treatment of surgical intervention
11. Use of tobacco, e-cigarette, nicotine, or marijuana products or significant history of drug or alcohol abuse within 6 months of screening.
12. Acute pulmonary embolism within 90 days of screening.
13. Participation in pulmonary rehabilitation within 90 days of screening.
14. Prior or concurrent use of any investigation drug/device/therapy or participation in any investigational study with therapeutic intent within 30 days or 5 half-lives, whichever is longer before the first dose of the IP.
15. BMI ≥40 kg/m2.
16. Uncontrolled hypertension as evidenced by systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg during the screening period. Subjects who fail screening due to high blood pressure can be re-screened once, after their antihypertensive medicines have been adjusted and doses have been stable for at least 4 weeks.
17. Concomitant disease that confers a life expectancy of <6 months at screening.
18. The Investigator judges that the subject will be unable to fully participate in the study and complete it for any reason, including inability to comply with the study procedures and treatment of addiction or any other relevant medical or psychiatric conditions.
19. High likelihood of lung transplantation (in the opinion of the Investigator) within 4 months after randomization.
20. History of liver dysfunction, including subjects with moderate (Child-Pugh B) or severe (Child Pugh C) impairment or disordered coagulation.
21. Female subjects who are pregnant or breastfeeding.
22. Worse than mild untreated sleep apnea (5-14.9 events/hour). Treated sleep apnea is permitted.

    Other Exclusions
23. History of allergic or anaphylactic reaction to mirivadelgat or to any component of the excipient.
24. Previous exposure to mirivadelgat.

    Diagnostic Assessments
25. The following laboratory parameters are excluded:

    * Hemoglobin <10 g/dL (100 g/L).
    * White blood cells (WBC) <3000/µL (<3000/mm3).
    * Platelet count <70,000/µL (70,000/mm3).
    * Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 or evidence of acute kidney injury.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Vascular Resistance (PVR) | 12 weeks
  The mean change from baseline to Week 12 in PVR assessed by right heart catheterization (RHC) for mirivadelgat vs. placebo.

SECONDARY OUTCOMES:
6-minute walk distance | 12 weeks
  The mean change from baseline to Week 12 in the 6-minute walk distance
Time to clinical deterioration from baseline to Week 12 for any of the following ADJUDICATED clinical events | 12 weeks
  * Death (all-cause mortality).
  * Hospital admission greater than 24 hours due to worsening of pulmonary hypertension.
  * Worsening of pulmonary hypertension resulting in the need for lung transplant or balloon atrial septostomy.
  * Initiation of parenteral prostanoid therapy, initiation of oxygen therapy, initiation of any other pulmonary hypertension-specific therapies, or need for an increase of diuretics for more than 4 weeks due to worsening of pulmonary hypertension.
  * Disease progression.
  * A decrease of more than 15% from the baseline in the 6-minute walk distance test combined with World Health Organization (WHO) functional class III or IV symptoms at 2 consecutive visits separated by at least 7 days.
Long-term prognostic risk factors | 12 weeks
  The mean change from baseline to Week 12 of long-term prognostic risk factors of plasma/serum N-terminal pro-brain natriuretic peptide (NT-ProBNP), C-terminal procollagen I (PICP), N-terminal procollagen I (NICP or PINP), and N-terminal procollagen III (NIIICP or PIIINP).
Patient-reported outcome measures (PROMS): (SF)-36v2 | 12 weeks
  The change from baseline to Week 12 in the Short Form (SF)-36v2 Health Survey with Scale 0 to 100 (mean is 50), 0 is worst, 100 is best
Patient-reported outcome measures (PROMS): WIQ | 12 weeks
  The change from baseline to Week 12 in the Walking Impairment Questionnaire (WIQ) with percentage scale ranging from 0% (worst) to 100% (best)
Patient-reported outcome measures (PROMS): PAH-SYMPACT | 12 weeks
  The change from baseline to Week 12 in the Pulmonary Arterial Hypertension-Symptoms and Impact Questionnaire (PAH-SYMPACT) with each point scored from 0 (best) to 4 (worst)

OTHER OUTCOMES:
Inflammatory markers | 12 weeks
  The mean change in concentration of inflammatory markers interleukin-6 (IL-6), high-sensitivity C-reactive protein (HS-CRP), and tumor necrosis factor- α (TNF-α) from baseline to Week 12.
Cardiac MRI fibrosis score | 12 weeks
  The mean change in cardiac MRI fibrosis score assessed by cardiac MRI gadolinium enhancement from baseline to Week 12 with a continuous variable that is not presented on a scale (only for subjects who have no contraindication to MRI procedure).
Quantitative ILD features | 12 weeks
  The change in Quantitative ILD features [i.e., Ground glass (QGC), Lung fibrosis (QLF), and Honeycombing (QHC)] assessed by HRCT scan from baseline to Week 12.
Risk for intervention | 12 weeks
  The Absolute Risk for intervention regarding specific events of death and stroke (CVA) (the absolute risk reduction between placebo and treatment of the composite event of death and stroke)
Cardiac strain | 12 weeks
  The mean change in cardiac strain assessed by contrast-enhancement echocardiogram from baseline to Week 12.
Change of right ventricle/left ventricle (RV/LV) size | 12 weeks
  The mean change in transthoracic echocardiography measurement of right ventricle/left ventricle (RV/LV) size, function, and strain from baseline to Week 12.
Pulmonary function tests (PFTs) - FEV1 | 12 weeks
  The change in FEV1 from baseline to Week 12.
Pulmonary function tests (PFTs) - FEV1 / FVC ratio | 12 weeks
  The change in FEV1 / FVC from baseline to Week 12.
Pharmacokinetic (PK) parameters: T1/2 | 12 weeks
  T1/2 for mirivadelgat and its active metabolite AD-835.
Pharmacokinetic (PK) parameters: AUC | 12 weeks
  AUC for mirivadelgat and its active metabolite AD-835.

CONTACTS AND LOCATIONS:
Overall Officials: Bassem Elmankabadi, MD, Study Director — Foresee Pharmaceuticals
Locations (9):
- Taiwan (9):
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan

IPD SHARING:
Plan to Share IPD: No